CLINICAL TRIAL: NCT04635423
Title: A Phase 3, Randomized, Placebo-controlled Clinical Study to Evaluate the Efficacy, Immunogenicity and Safety of the 9vHPV Vaccine in Japanese Males, 16 to 26 Years of Age.
Brief Title: Efficacy, Immunogenicity, and Safety Study of the 9vHPV Vaccine in Japanese Males (V503-064)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V503-064; V503-064 (Other: MSD Protocol Number); jRCT2031200217 (Registry Identifier: jRCT); 2020-001047-67 (EudraCT Number)
Record Dates: First submitted 2020-11-05; First posted 2020-11-19 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Warts, Genital; Neoplasms, Anal
MeSH Terms: conditions — Condylomata Acuminata; Anus Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V503 (Experimental): Participants receive an intramuscular (IM) injection of V503 (9-valent human papillomavirus [9vHPV] vaccine) at Day 1, Month 2, and Month 6.
  Interventions: Biological: V503
- Placebo (Placebo Comparator): Participants receive an IM injection of placebo at Day 1, Month 2, and Month 6.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: V503 — 9-valent vaccine, HPV 6/11/16/18/31/33/45/52/58, L1 virus-like particle (VLP) 30/40/60/40/20/20/20/20/20 mcg per dose.
  Other Names: 9vHPV vaccine; SILGARD®9; GARDASIL™9
  Arms: V503
Other: Placebo — 0.9% sodium chloride (NaCL)
  Arms: Placebo

SUMMARY:
The purposes of this phase 3, double-blind, placebo-controlled clinical study are to evaluate the efficacy of V503 (9-valent human papillomavirus [9vHPV] vaccine) in preventing human papillomavirus (HPV)-related anogenital persistent infection, and to evaluate the safety/tolerability of V503, in Japanese males who are 16 to 26 years of age. It is hypothesized that administration of a 3-dose regimen of V503 reduces the combined incidence of HPV 6/11/16/18-related anogenital persistent infection, as well as the combined incidence of HPV 31/33/45/52/58-related anogenital persistent infection, compared with placebo.

The study includes a Base Study to assess efficacy and safety of V503, and an Extension Study. Participants who received placebo in the Base Study will be eligible to receive V503 vaccine on Day 1, Month 2, and Month 6 of the Extension Study. Participants who received less than 3 doses of V503 in the Base Study will be offered the opportunity to complete the 3-dose regimen in the Extension Study.

ELIGIBILITY:
Inclusion Criteria:

* Is a Japanese male 16 to 26 years of age
* Has no more than 5 lifetime sexual partners

Exclusion Criteria:

* Has a history of known prior vaccination with an HPV vaccine or plans to receive one outside the study
* Has a history of external genital warts
* Has a history of severe allergic reaction that required medical intervention
* Has received immune globulin or blood-derived products in the past 3 months or plan to receive any before Month 7 of the study
* Has a history of splenectomy, is currently immunocompromised, or has been diagnosed with immunodeficiency, human immunodeficiency virus (HIV), lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition
* Has received immunosuppressive therapy in the past year, excluding inhaled, nasal, or topical corticosteroids and certain regimens of systemic corticosteroids
* Has a known thrombocytopenia or coagulation disorder that would contraindicate intramuscular injections
* Has ongoing alcohol or drug abuse within the past 12 months

Ages: 16 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 1059 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (22):
- Japan (22):
  - Umeyama Clinic ( Site 6406), Takasaki, Gunma
  - Association of Healthcare Corporation Koukankai Koukan Clinic ( Site 6424), Kawasaki, Kanagawa
  - Ocean Clinic ( Site 6407), Yokohama, Kanagawa
  - Kanno Clinic ( Site 6402), Sakai, Osaka
  - P-One Clinic, Keikokai Medical Corp. ( Site 6419), Hachiōji, Tokyo
  - Iwasa Clinic ( Site 6411), Osaka
  - Nomura Clinic Namba ( Site 6405), Osaka
  - Medical Corporation Seiwakai Hayakawa Clinic ( Site 6409), Osaka
  - Yamanaka Clinic ( Site 6410), Osaka
  - Doujin Memorial Medical Foundation, Meiwa Hospital ( Site 6404), Tokyo
  - Yuge Clinic ( Site 6421), Tokyo
  - Taisei Clinic ( Site 6403), Tokyo
  - Mildix Skin Clinic ( Site 6423), Tokyo
  - Sugisawa Dermatology Clinic ( Site 6422), Tokyo
  - Medical Corporation Sanshikai Toru Clinic ( Site 6401), Tokyo
  - Medical Corporation Mori to Umi Tokyo Tokyo Kamata Hospital ( Site 6418), Tokyo
  - Seiyukai Medical Corporation Itoh Skin Clinic ( Site 6416), Tokyo
  - Naoko Dermatology Clinic ( Site 6417), Tokyo
  - Medical Corporation Iseikai My City Clinic ( Site 6414), Tokyo
  - Shinjuku Higashiguchi Clinic ( Site 6415), Tokyo
  - Ogikuboekimae Clinic ( Site 6413), Tokyo
  - Kusunoki Clinic ( Site 6412), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | V503 | Placebo
Started | 529 | 530
Vaccination 1: Day 1 | 529 | 530
Vaccination 2: Month 2 | 523 | 518
Vaccination 3: Month 6 | 514 | 508
Completed | 0 | 0
Not Completed | 529 | 530
Not completed — Ongoing | 493 | 501
Not completed — Withdrawal by Subject | 36 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V503 | Placebo | Total
Number analyzed (Participants) | 529 | 530 | 1059
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.9 (2.1) | 22.8 (2.1) | 22.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 529 | 530 | 1059
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 529 | 530 | 1059
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 529 | 530 | 1059
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Sexual Orientation Participant Subgroups [Count of Participants; unit: Participants] — Participant randomization was stratified by sexual orientation heterosexual males (HM) or males who have sex with males (MSM). For HM, participants must be a heterosexual male, who has had exclusively female sexual partners, and has 1 to 5 lifetime female sexual partners at the time of enrollment. For MSM, participants must identify themselves as a male who has sex with males, must have engaged in either anal intercourse or oral sex with another male sexual partner within the last year, and have 0 to 5 lifetime male and/or female sexual partners at the time of enrollment.
  Participants
    Heterosexual Males (HM) | 473 | 474 | 947
    Males Who Have Sex With Males (MSM) | 56 | 56 | 112

OUTCOME MEASURES:

1. Primary Outcome: Combined Incidence of Human Papillomavirus (HPV) 6/11/16/18-related Anogenital Persistent Infection
Description: Combined incidence of HPV type(s) 6/11/16/18-related anogenital persistent infection was defined to have occurred in a participant; 1) who is polymerase chain reaction (PCR) positive to at least one applicable HPV type(s) in 2 consecutive anogenital or biopsy samples from at least 2 consecutive visits 6 months (±1 month visit) or longer apart, or 2) who has a pathology diagnosis of condyloma, penile/perineal/perianal intraepithelial neoplasia, or penile, perineal or perianal cancer and PCR detection of at least one applicable HPV type(s) in an adjacent section and PCR positive for the same HPV type at a separate adjacent visit with regardless of visit interval, prior to or following the biopsy showing HPV disease. Incidence was defined as the number of cases per 100 person-years of follow-up in both V503 and placebo arms. Per protocol, cases per 100 person-years is reported for applicable HPV type eligible participants with data available in the per-protocol efficacy population (PPE).
Time Frame: Up to approximately 36 Months
Population: HPV type 6/11/16/18 eligible participants with data available in PPE population within acceptable day ranges; received all 3 vaccinations of correct dose within 1 year, Month 7 swab samples collected postdose 3 with PCR result, seronegative to the appropriate HPV type at baseline and PCR-negative to appropriate HPV type on all samples collected from baseline through Month 7, and no protocol deviations that could interfere with the evaluation of participant's immune response to the 9vHPV vaccine.
Measure: Number; unit: Cases per 100 Person-years
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 496 | 483
Cases per 100 Person-years | 0.2 | 2.2
Statistical Analysis 1: Comparison: V503 vs Placebo; Test type: Superiority; p < 0.001, Exact Binomial Method Chan and Bohidar — one-sided p-value based on exact binomial method proposed by Chan and Bohidar; Observed Efficacy (%) = 89.3, 95% CI 2-sided [55.4 to 98.2] — The statistical criterion for success requires that the lower bound of the 2-sided 95% confidence interval (CI) for vaccine efficacy (VE) against the primary efficacy endpoint is greater than 0%

2. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The participant recorded the presence of any vaccination report card (VRC)-prompted injection-site AEs that occurred in the 5 days after any vaccination. The percentage of participants with an injection-site AE prompted on the VRC (redness/erythema, tenderness/pain, and swelling) is reported here for all randomized participants in the All Participants as Treated (APaT) population.
Time Frame: Up to 5 days after any vaccination
Population: All Participants as Treated (APaT) population, all randomized participants who received at least 1 dose of the V503 vaccine or placebo and have provided safety data at any time during the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 529 | 530
Percentage of Participants | 69.8 | 29.6
Statistical Analysis 1: Comparison: V503 vs Placebo; Test type: Other; Miettinen & Nurminen method; Difference in Percentages = 40.1, 95% CI 2-sided [34.5 to 45.5] — Difference in percentages calculated as % V503 minus % Placebo

3. Primary Outcome: Percentage of Participants With ≥1 Systemic AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least 1 systemic AE is reported here for all randomized participants in the All Participants as Treated (APaT) population.
Time Frame: Up to 15 days after any vaccination
Population: All Participants as Treated (APaT) population, which consists of all randomized participants who received at least 1 dose of the V503 vaccine or placebo and have provided safety data at any time during the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 529 | 530
Percentage of Participants | 20.2 | 19.8
Statistical Analysis 1: Comparison: V503 vs Placebo; Test type: Other; Miettinen & Nurminen method; Difference in Percentage = 0.4, 95% CI 2-sided [-4.4 to 5.2] — Difference in percentages calculated as % V503 minus % Placebo

4. Primary Outcome: Percentage of Participants With ≥1 Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention, that results in death, is life-threatening, requires hospitalization or prolongs existing hospitalization, results in persistent/significant disability/incapacity, is a congenital birth defect, or is another important medical event. The percentage of participants who experienced at least 1 SAE is reported here for all randomized participants in the All Participants as Treated (APaT) population.
Time Frame: Up to approximately 37 months
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 529 | 530
Percentage of Participants | 1.3 | 0.9

5. Primary Outcome: Number of Participants With Elevated Oral Body Temperature
Description: Participants collected their oral body temperature in the evening of their vaccination day and at the same time each day thereafter for 4 days. The maximum body temperature obtained within 5 days of any of the 3 vaccinations was recorded using the vaccination report card (VRC). Per protocol, fever was defined as an oral temperature of ≥99.5°F(37.5°C). The number of participants who had at least 1 oral body temperature reading that was, <99.5°F (<37.5ºC), ≥99.5°F (≥37.5ºC) and <100.4°F (38.0°C), or ≥100.4°F (38.0°C) and <101.3°F(38.5°C), or ≥101.3°F(38.5°C) is reported here for all randomized participants in the APaT population with temperature data available.
Time Frame: Up to 5 days after any vaccination
Population: All Participants as Treated (APaT) population with temperature data available. APaT consists of all randomized participants who received at least 1 dose of the V503 vaccine or placebo and have provided safety data at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 527 | 526
Participants
  <99.5°F (37.5°C) | 502 | 496
  ≥99.5°F (≥37.5ºC) and <100.4°F (38.0°C) | 19 | 22
  ≥100.4°F (38.0°C) and <101.3°F(38.5°C) | 1 | 1
  ≥101.3°F(38.5°C) | 5 | 7

6. Secondary Outcome: Combined Incidence of HPV 31/33/45/52/58-related Anogenital Persistent Infection
Description: Combined incidence of HPV type(s) 31/33/45/52/58-related anogenital persistent infection was defined to have occurred in a participant; 1) who is polymerase chain reaction (PCR) positive to at least 1 applicable HPV type(s) in 2 consecutive anogenital or biopsy samples from at least 2 consecutive visits 6 months (±1 month visit) or longer apart, or 2) who has a pathology diagnosis of condyloma, penile/perineal/perianal intraepithelial neoplasia, or penile, perineal or perianal cancer and PCR detection of at least 1 applicable HPV type in an adjacent section and PCR positive for the same HPV type at a separate adjacent visit with regardless of visit interval, prior to or following the biopsy showing HPV disease. Incidence was defined as the number of cases per 100 person-years of follow-up in both V503 and placebo arms. Per protocol, cases per 100 person-years is reported for applicable HPV type(s) eligible participants with data available in the per-protocol efficacy population (PPE).
Time Frame: Up to approximately 36 Months
Population: HPV type 31/33/45/52/58 eligible participants with data available in PPE population within acceptable day ranges; received all 3 vaccinations of correct dose within 1 year, Month 7 swab samples collected postdose 3 with PCR result, seronegative to appropriate HPV type at baseline and PCR-negative to appropriate HPV type on all samples collected from baseline through Month 7, and no protocol deviations that could interfere with the evaluation of participant's immune response to the 9vHPV vaccine.
Measure: Number; unit: cases per 100 Person-years
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 505 | 493
cases per 100 Person-years | 0.7 | 1.9
Statistical Analysis 1: Comparison: V503 vs Placebo; Test type: Superiority; p = 0.023, Exact Binomial Method Chan and Bohidar — one-sided p-value based on exact binomial method proposed by Chan and Bohidar; Observed Efficacy (%) = 63.5, 95% CI 2-sided [2.7 to 86.0] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV 6/11/16/18/31/33/45/52/58 - All Randomized Participants
Description: Antibodies to the HPV types 6/11/16/18/31/33/45/52/58 contained in V503 were measured using a competitive Luminex immunoassay (cLIA). Per protocol, antibody titers were expressed as milli Merck units/milliliter (mMU/mL). Geometric Mean Titers (GMTs) is reported for both V503 and Placebo for all randomized participants of the per-protocol immunogenicity population (PPI).
Time Frame: Month 7
Population: Eligible all randomized participants PPI population; within acceptable day ranges; received 3 vaccinations of correct dose within 1 year, Month 7 swab samples collected postdose 3 with PCR result, seronegative to appropriate HPV type(s) at baseline and PCR-negative to appropriate HPV type(s) on samples collected from baseline through Month 7, provided serological samples, and had no protocol deviations that could interfere with the evaluation of participant's immune response to the V503 vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 456 | 458
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 399 | 367
  Anti-HPV 6 | 927.3 [850.2 to 1011.3] | 21.1 [NA to 22.5] — NA: < Lower Limit of Quantification (LLOQ) of 20 mMU/mL
  Anti-HPV 11: number analyzed (Participants) | 399 | 367
  Anti-HPV 11 | 716.5 [654.4 to 784.5] | NA [NA to NA] — NA: < LLOQ of 16 mMU/mL
  Anti-HPV 16: number analyzed (Participants) | 449 | 446
  Anti-HPV 16 | 3491.6 [3196.5 to 3814.0] | NA [NA to NA] — NA: < LLOQ of 20 mMU/mL
  Anti-HPV 18: number analyzed (Participants) | 417 | 411
  Anti-HPV 18 | 998.0 [904.3 to 1101.4] | 45.5 [43.4 to 47.7]
  HPV-31: number analyzed (Participants) | 435 | 429
  HPV-31 | 832.1 [753.3 to 919.2] | 15.4 [14.3 to 16.5]
  HPV-33: number analyzed (Participants) | 451 | 442
  HPV-33 | 489.8 [448.6 to 534.7] | 12.7 [11.9 to 13.4]
  Anti-HPV 45: number analyzed (Participants) | 439 | 434
  Anti-HPV 45 | 326.6 [293.7 to 363.2] | 8.5 [NA to 9.0] — NA: < LLOQ of 8 mMU/mL
  Anti-HPV 52: number analyzed (Participants) | 437 | 433
  Anti-HPV 52 | 390.5 [356.3 to 428.0] | 10.1 [9.5 to 10.8]
  Anti-HPV 58 | 588.3 [537.7 to 643.6] | NA [NA to NA] — NA: < LLOQ of 8 mMU/mL

8. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV 6/11/16/18/31/33/45/52/58 - Heterosexual Males (HM) Participant Subgroup
Description: Antibodies to the HPV types 6/11/16/18/31/33/45/52/58 contained in V503 were measured using a competitive Luminex immunoassay (cLIA). Per protocol, antibody titers were expressed as milli Merck units/milliliter (mMU/mL). Geometric Mean Titers (GMTs) is reported for both V503 and Placebo for the heterosexual males (HM) subgroup of the per-protocol immunogenicity population (PPI).
Time Frame: Month 7
Population: HM subgroup of the PPI population; within the acceptable day ranges, received 3 vaccinations of correct dose within 1 year, Month 7 swab samples collected postdose 3 with PCR result, seronegative to appropriate HPV type(s) at baseline and PCR-negative to appropriate HPV type(s) on all samples collected from baseline through Month 7, provided serological samples, and had no protocol deviations that could interfere with the evaluation of participant's immune response to the V503 vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 408 | 415
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 360 | 339
  Anti-HPV 6 | 950.2 [866.8 to 1041.6] | 21.0 [NA to 22.6] — NA: < Lower Limit of Quantitation (LLOQ) of 20 mMU/mL
  Anti-HPV 11: number analyzed (Participants) | 360 | 339
  Anti-HPV 11 | 730.6 [664.4 to 803.4] | NA [NA to NA] — NA: < LLOQ of 16 mMU/mL
  Anti-HPV 16: number analyzed (Participants) | 404 | 404
  Anti-HPV 16 | 3608.3 [3288.6 to 3959.0] | NA [NA to NA] — NA: < LLOQ of 20 mMU/mL
  Anti-HPV 18: number analyzed (Participants) | 373 | 369
  Anti-HPV 18 | 1044.7 [942.7 to 1157.7] | 45.1 [42.9 to 47.3]
  Anti-HPV 31: number analyzed (Participants) | 387 | 384
  Anti-HPV 31 | 867.8 [780.7 to 964.7] | 15.1 [14.0 to 16.3]
  Anti-HPV 33: number analyzed (Participants) | 404 | 396
  Anti-HPV 33 | 495.4 [451.9 to 543.1] | 12.6 [11.8 to 13.4]
  Anti-HPV 45: number analyzed (Participants) | 396 | 389
  Anti-HPV 45 | 333.8 [298.4 to 373.5] | 8.4 [NA to 9.0] — NA: < LLOQ of 8 mMU/mL
  Ant-HPV 52: number analyzed (Participants) | 392 | 390
  Ant-HPV 52 | 408.7 [372.1 to 448.9] | 10.0 [9.3 to 10.7]
  Anti-HPV 58 | 609.1 [554.2 to 669.4] | NA [NA to NA] — NA: < LLOQ of 8 mMU/mL

9. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV 6/11/16/18/31/33/45/52/58 - Males Who Have Sex With Males (MSM) Participant Subgroup
Description: Antibodies to the HPV types 6/11/16/18/31/33/45/52/58 contained in V503 were measured using a competitive Luminex immunoassay (cLIA). Per protocol, antibody titers were expressed as milli Merck units/milliliter (mMU/mL). Geometric Mean Titers (GMTs) is reported for both V503 and Placebo for the males who have sex with males (MSM) subgroup of the per-protocol immunogenicity population (PPI).
Time Frame: Month 7
Population: MSM subgroup of the PPI population; within the acceptable day ranges, received 3 vaccinations of correct dose within 1 year, Month 7 swab samples collected postdose 3 with PCR result, seronegative to appropriate HPV type(s) at baseline and PCR-negative to appropriate HPV type(s) on all samples collected from baseline through Month 7, provided serological samples, and had no protocol deviations that could interfere with the evaluation of participant's immune response to the V503 vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 48 | 46
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 39 | 28
  Anti-HPV 6 | 740.2 [569.2 to 962.6] | 21.5 [NA to 27.5] — NA: < Lower Limit of Quantification (LLOQ) of 20 mMU/mL
  Anti-HPV 11: number analyzed (Participants) | 39 | 28
  Anti-HPV 11 | 598.8 [438.7 to 817.3] | NA [NA to NA] — NA: < LLOQ of 16 mMU/mL
  Anti-HPV 16: number analyzed (Participants) | 45 | 42
  Anti-HPV 16 | 2599.5 [1957.4 to 3452.4] | NA [NA to NA] — NA: < LLOQ of 20 mMU/mL
  Anti-HPV 18: number analyzed (Participants) | 44 | 42
  Anti-HPV 18 | 677.4 [487.6 to 941.0] | 49.7 [42.1 to 58.6]
  Anti-HPV 31: number analyzed (Participants) | 48 | 45
  Anti-HPV 31 | 593.2 [446.0 to 789.0] | 17.7 [14.1 to 22.2]
  Anti-HPV 33: number analyzed (Participants) | 47 | 46
  Anti-HPV 33 | 443.6 [327.9 to 600.1] | 13.5 [11.5 to 16.0]
  Anti-HPV 45: number analyzed (Participants) | 43 | 45
  Anti-HPV 45 | 266.6 [190.1 to 373.8] | 9.1 [NA to 11.1] — NA: < LLOQ of 8 mMU/mL
  Anti-HPV 52: number analyzed (Participants) | 45 | 43
  Anti-HPV 52 | 262.9 [186.7 to 370.2] | 11.3 [9.0 to 14.2]
  Anti-HPV 58: number analyzed (Participants) | 48 | 43
  Anti-HPV 58 | 437.7 [327.8 to 584.5] | NA [NA to 8.4] — NA: < LLOQ of 8 mMU/mL

10. Secondary Outcome: Percentage of Participants With Seroconversion to HPV 6/11/16/18/31/33/45/52/58 - All Randomized Participants
Description: Percentage of seroconversion to each of HPV 6/11/16/18/31/33/45/52/58 at Month 7 based on competitive Luminex immunoassay (cLIA) from participant serum samples. Seroconversion is defined as changing a participant's serostatus from seronegative at Day 1 to seropositive at 1 month post last dose Month 7. A participant with anti-HPV cLIA titer at or above the serostatus cutoff values of the cLIA for a given HPV type is considered seropositive for that HPV type. The serostatus cutoffs (milli Merck units/milliliter (mMU/mL)) for HPV types were as follows: HPV Type 6: ≥65, HPV Type 11: ≥37; HPV Type 16: ≥79, HPV Type 18: ≥85, HPV Type 31: ≥46, HPV Type 33: ≥26, HPV Type 45: ≥21, HPV Type 52: ≥30, and HPV Type 58: ≥31. The percentage of participants with seroconversion is reported for both V503 and Placebo for all randomized participants of the per-protocol immunogenicity population (PPI).
Time Frame: Month 7
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 456 | 458
Percentage of Participants
  Anti-HPV 6 cLIA ≥65 mMU/mL: number analyzed (Participants) | 399 | 367
  Anti-HPV 6 cLIA ≥65 mMU/mL | 99.7 [98.6 to 100.0] | 3.5 [1.9 to 6.0]
  Anti-HPV 11 cLIA ≥37 mMU/mL: number analyzed (Participants) | 399 | 367
  Anti-HPV 11 cLIA ≥37 mMU/mL | 99.7 [98.6 to 100.0] | 4.1 [2.3 to 6.7]
  Anti-HPV 16 cLIA ≥79 mMU/mL: number analyzed (Participants) | 449 | 446
  Anti-HPV 16 cLIA ≥79 mMU/mL | 99.6 [98.4 to 99.9] | 4.3 [2.6 to 6.6]
  Anti-HPV 18 cLIA ≥85 mMU/mL: number analyzed (Participants) | 417 | 411
  Anti-HPV 18 cLIA ≥85 mMU/mL | 99.3 [97.9 to 99.9] | 8.3 [5.8 to 11.4]
  Anti-HPV 31 cLIA ≥46 mMU/mL: number analyzed (Participants) | 435 | 429
  Anti-HPV 31 cLIA ≥46 mMU/mL | 98.9 [97.3 to 99.6] | 5.6 [3.6 to 8.2]
  Anti-HPV 33 cLIA ≥26 mMU/mL: number analyzed (Participants) | 451 | 442
  Anti-HPV 33 cLIA ≥26 mMU/mL | 99.8 [98.8 to 100.0] | 11.1 [8.3 to 14.4]
  Anti-HPV 45 cLIA ≥21 mMU/mL: number analyzed (Participants) | 439 | 434
  Anti-HPV 45 cLIA ≥21 mMU/mL | 98.9 [97.4 to 99.6] | 9.0 [6.5 to 12.1]
  Anti-HPV 52 cLIA ≥30 mMU/mL: number analyzed (Participants) | 437 | 433
  Anti-HPV 52 cLIA ≥30 mMU/mL | 98.9 [97.4 to 99.6] | 4.2 [2.5 to 6.5]
  Anti-HPV 58 cLIA ≥31 mMU/mL | 99.3 [98.1 to 99.9] | 1.5 [0.6 to 3.1]

11. Secondary Outcome: Percentage of Participants With Seroconversion to HPV 6/11/16/18/31/33/45/52/58 - Heterosexual Males (HM) Participant Subgroup
Description: Percentage of seroconversion to each of HPV 6/11/16/18/31/33/45/52/58 at Month 7 based on competitive Luminex immunoassay (cLIA) from participant serum samples. Seroconversion is defined as changing a participant's serostatus from seronegative at Day 1 to seropositive at 1 month post last dose Month 7. A participant with anti-HPV cLIA titer at or above the serostatus cutoff values of the cLIA for a given HPV type is considered seropositive for that HPV type. The serostatus cutoffs (milli Merck units/milliliter (mMU/mL)) for HPV types were as follows: HPV Type 6: ≥65, HPV Type 11: ≥37; HPV Type 16: ≥79, HPV Type 18: ≥85, HPV Type 31: ≥46, HPV Type 33: ≥26, HPV Type 45: ≥21, HPV Type 52: ≥30, and HPV Type 58: ≥31. The percentage of participants with seroconversion is reported for both V503 and Placebo for the heterosexual males (HM) subgroup of the per-protocol immunogenicity population (PPI).
Time Frame: Month 7
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 408 | 415
Percentage of Participants
  Anti-HPV 6 cLIA ≥65 mMU/mL: number analyzed (Participants) | 360 | 339
  Anti-HPV 6 cLIA ≥65 mMU/mL | 99.7 [98.5 to 100.0] | 3.5 [1.8 to 6.1]
  Anti-HPV 11 cLIA ≥37 mMU/mL: number analyzed (Participants) | 360 | 339
  Anti-HPV 11 cLIA ≥37 mMU/mL | 99.7 [98.5 to 100.0] | 4.4 [2.5 to 7.2]
  Anti-HPV 16 cLIA ≥79 mMU/mL: number analyzed (Participants) | 404 | 404
  Anti-HPV 16 cLIA ≥79 mMU/mL | 99.5 [98.2 to 99.9] | 3.7 [2.1 to 6.0]
  Anti-HPV 18 cLIA ≥85 mMU/mL: number analyzed (Participants) | 373 | 369
  Anti-HPV 18 cLIA ≥85 mMU/mL | 99.5 [98.1 to 99.9] | 7.6 [5.1 to 10.8]
  Anti-HPV 31 cLIA ≥46 mMU/mL: number analyzed (Participants) | 387 | 384
  Anti-HPV 31 cLIA ≥46 mMU/mL | 99.0 [97.4 to 99.7] | 5.2 [3.2 to 7.9]
  Anti-HPV 33 cLIA ≥26 mMU/mL: number analyzed (Participants) | 404 | 396
  Anti-HPV 33 cLIA ≥26 mMU/mL | 99.8 [98.6 to 100.0] | 11.4 [8.4 to 14.9]
  Anti-HPV 45 cLIA ≥21 mMU/mL: number analyzed (Participants) | 396 | 389
  Anti-HPV 45 cLIA ≥21 mMU/mL | 98.7 [97.1 to 99.6] | 8.5 [5.9 to 11.7]
  Anti-HPV 52 cLIA ≥30 mMU/mL: number analyzed (Participants) | 392 | 390
  Anti-HPV 52 cLIA ≥30 mMU/mL | 99.2 [97.8 to 99.8] | 3.8 [2.2 to 6.3]
  Anti-HPV 58 cLIA ≥31 mMU/mL | 99.3 [97.9 to 99.8] | 1.7 [0.7 to 3.4]

12. Secondary Outcome: Percentage of Participants With Seroconversion to HPV 6/11/16/18/31/33/45/52/58 - Males Who Have Sex With Males (MSM) Participant Subgroup
Description: Percentage of seroconversion to each of HPV 6/11/16/18/31/33/45/52/58 at Month 7 based on competitive Luminex immunoassay (cLIA) from participant serum samples. Seroconversion is defined as changing a participant's serostatus from seronegative at Day 1 to seropositive at 1 month post last dose Month 7. A participant with anti-HPV cLIA titer at or above the serostatus cutoff values of the cLIA for a given HPV type is considered seropositive for that HPV type. The serostatus cutoffs (milli Merck units/milliliter (mMU/mL)) for HPV types were as follows: HPV Type 6: ≥65, HPV Type 11: ≥37; HPV Type 16: ≥79, HPV Type 18: ≥85, HPV Type 31: ≥46, HPV Type 33: ≥26, HPV Type 45: ≥21, HPV Type 52: ≥30, and HPV Type 58: ≥31. The percentage of participants with seroconversion is reported for both V503 and Placebo for the males who have sex with males (MSM) subgroup of the per-protocol immunogenicity population (PPI).
Time Frame: Month 7
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V503 | Placebo
Number analyzed (Participants) | 48 | 46
Percentage of Participants
  Anti-HPV 6 cLIA ≥65 mMU/mL: number analyzed (Participants) | 39 | 28
  Anti-HPV 6 cLIA ≥65 mMU/mL | 100.0 [91.0 to 100.0] | 3.6 [0.1 to 18.3]
  Anti-HPV 11 cLIA ≥37 mMU/mL: number analyzed (Participants) | 39 | 28
  Anti-HPV 11 cLIA ≥37 mMU/mL | 100.0 [91.0 to 100.0] | 0.0 [0.0 to 12.3]
  Anti-HPV 16 cLIA ≥79 mMU/mL: number analyzed (Participants) | 45 | 42
  Anti-HPV 16 cLIA ≥79 mMU/mL | 100.0 [92.1 to 100.0] | 9.5 [2.7 to 22.6]
  Anti-HPV 18 cLIA ≥85 mMU/mL: number analyzed (Participants) | 44 | 42
  Anti-HPV 18 cLIA ≥85 mMU/mL | 97.7 [88.0 to 99.9] | 14.3 [5.4 to 28.5]
  Anti-HPV 31 cLIA ≥46 mMU/mL: number analyzed (Participants) | 48 | 45
  Anti-HPV 31 cLIA ≥46 mMU/mL | 97.9 [88.9 to 99.9] | 8.9 [2.5 to 21.2]
  Anti-HPV 33 cLIA ≥26 mMU/mL: number analyzed (Participants) | 47 | 46
  Anti-HPV 33 cLIA ≥26 mMU/mL | 100.0 [92.5 to 100.0] | 8.7 [2.4 to 20.8]
  Anti-HPV 45 cLIA ≥21 mMU/mL: number analyzed (Participants) | 43 | 45
  Anti-HPV 45 cLIA ≥21 mMU/mL | 100.0 [91.8 to 100.0] | 13.3 [5.1 to 26.8]
  Anti-HPV 52 cLIA ≥30 mMU/mL: number analyzed (Participants) | 45 | 43
  Anti-HPV 52 cLIA ≥30 mMU/mL | 95.6 [84.9 to 99.5] | 7.0 [1.5 to 19.1]
  Anti-HPV 58 cLIA ≥31 mMU/mL: number analyzed (Participants) | 48 | 43
  Anti-HPV 58 cLIA ≥31 mMU/mL | 100.0 [92.6 to 100.0] | 0.0 [0.0 to 8.2]

ADVERSE EVENTS:
Time Frame: Up to approximately 37 months
Description: Population for All-cause mortality was All Randomized Participants. Population for Non-serious adverse events and serious adverse events was All Participants as Treated (APaT). The APaT population consists of all randomized participants who received at least 1 dose of the V503 (9vHPV) vaccine or placebo and have provided safety data at any time during the study.
Arm/Group | V503 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/529 | 0/530
Serious Adverse Events (participants affected / at risk) | 7/529 | 5/530
Other Adverse Events (participants affected / at risk) | 374/529 | 183/530
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V503 (N=529) | Placebo (N=530)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V503 (N=529) | Placebo (N=530)
Injection site erythema (General disorders) | 104 (149) | 70 (101)
Injection site pain (General disorders) | 360 (739) | 122 (166)
Injection site swelling (General disorders) | 118 (164) | 40 (50)
Pyrexia (General disorders) | 29 (35) | 33 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT04635423/Prot_SAP_000.pdf